CLINICAL TRIAL: NCT00749047
Title: A Study on the Anti-proteinuric Effects of Pioglitazone in Patients With Type 2 Diabetes.
Brief Title: How Does the Diabetes Drug, Pioglitazone, Reduce Protein Loss in the Urine?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Christchurch Hospital (Other)
Responsible Party: Dr Brett Shand, Lipid and Diabetes Research Group, Christchurch Hospital, New Zealand.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H6E-AY-O017
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pioglitazone; Open study; Proteinuria; Glomerular selectivity indices
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Open label arm
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 15-45 mg/day
  Other Names: Actos; Batch number A490463

SUMMARY:
Pioglitazone is an insulin sensitising drug used in the treatment of patients with type 2 diabetes. In addition to its blood sugar lowering effect, pioglitazone also has a number of other beneficial effects, one of which is to reduce the loss of protein in the urine. The mechanism of this protein "sparing effect" of pioglitazone is not fully understood. The proposed study will investigate whether pioglitazone has beneficial effects on the filtration characteristics of filters in the kidney that are responsible for retaining protein in the body. The effect of pioglitazone on the size of the pores in the filters and also the electrostatic charge barriers that surround these pores will be investigated. The clinical study will involve 12 patients with type 2 diabetes with minimal urine protein loss, taking low dose pioglitazone for 3 months. Blood and urine samples will be collected at the beginning, mid point and end of the study and used to measure the concentration of specific proteins of different size and electrostatic charge. This data will be used to identify and characterise changes in the filtration properties of the kidney filters during the study.

DETAILED DESCRIPTION:
In addition to their insulin sensitising action, thiazolidinediones (TZDs) have beneficial effects on vascular function. These include a decrease in proteinuria and amelioration of diabetic nephropathy. Although the anti-proteinuric effect of TZDs is well established the mechanism(s) underlying these changes has yet to be determined. Possible mechanisms include altered renal haemodynamics, maintenance of anionic electrostatic filtration barriers in the glomerular basement membrane and pleiotropic effects.

The target of TZDs, the peroxisome proliferator-activated receptors (PPARs), directly modulate vessel wall function. The kidney differentially expresses all PPAR isoforms and there is evidence that TZDs have pleiotropic effects in the kidney over and above their metabolic and haemodynamic actions. These effects include a direct action on cultured mesangial cells, inhibition of in vivo mesangial expansion, reduction in podocyte injury, and decreased production of type IV collagen and urinary endothelin-1 levels in early stage diabetic nephropathy.

Glomerular ultrafiltration of plasma proteins is governed by the size of the filtration pores and the extent of anionic sites in the basement membrane and podocyte slit pore junction. It is possible that the anti-proteinuric effect of TZDs is attributable to an increase in size and/or charge selectivity in the glomerular filtration barrier. A Medline search showed there have been no studies on the effect of TZDs on protein ultrafiltration. The aim of the proposed study is to measure urinary protein size and charge selectivity in patients with early stage diabetic nephropathy before and after treatment with the TZD, pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, Type 2
* Age 18-70 yrs

Exclusion Criteria:

* Overt proteinuria (urine albumin:creatinine ratio >10.0
* Plasma creatinine 0.15 mmol/L
* HbA1c >10%
* Hear failure Class III or IV
* Peripheral oedema
* Abnormal liver function (serum AST >2.5 times upper limit of normal)
* Pregnancy or breastfeeding
* History of urinary tract infections
* Serious concomitant disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in proteinuria | 3 months

SECONDARY OUTCOMES:
Reduction in non-fasting plasma glucose concentration | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Christchurch Hospital, Christchurch, Canterbury, New Zealand